CLINICAL TRIAL: NCT06862947
Title: Effects of Preoperative Bilateral Rectus Sheath Block Guided by Ultrasound on Analgesic Efficacy and Recovery in Gynecological Single-Port Laparoscopy: A Prospective Randomized Double-Blind Placebo-Controlled Study
Brief Title: Ultrasound-Guided Rectus Sheath Block in Gynecological Single-Port Laparoscopy
Acronym: RSB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Jinjiang Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Fei Jia, Director of Anesthesiology Department, Chengdu Jinjiang Maternity and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202214
Record Dates: First submitted 2025-02-27; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Gynecological Laparoscopy; Postoperative Pain; Rectus Sheath Block
Keywords: Gynecology; Single-Port Laparoscopy; Rectus Sheath Block; Postop Pain Management
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was designed as a double-blind trial, ensuring that neither the patients nor the operating surgeons were aware of the group allocations throughout the study. This blinding was critical to eliminate bias in treatment administration and outcome assessment, thereby enhancing the validity of the trial results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-Guided Rectus Sheath Block (Active Comparator): Participants receive bilateral rectus sheath block with 15 ml of 0.4% ropivacaine on each side under ultrasound guidance
  Interventions: Procedure: Rectus Sheath Block
- Placebo (Placebo Comparator): articipants receive an equal volume of 0.9% saline as a placebo
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Rectus Sheath Block — Bilateral rectus sheath block performed under ultrasound guidance using 15 ml of 0.4% ropivacaine on each side
  Arms: Ultrasound-Guided Rectus Sheath Block
Procedure: Placebo — Injection of 15 ml of 0.9% saline as a placebo under the same conditions as the experimental group.
  Arms: Placebo

SUMMARY:
Title: Ultrasound-Guided Rectus Sheath Block in Gynecological Single-Port Laparoscopy

Brief Summary:

This study aims to evaluate the effects of preoperative ultrasound-guided bilateral rectus sheath block (RSB) on analgesic efficacy and recovery outcomes in patients undergoing gynecological single-port laparoscopy. The study is a prospective, randomized, double-blind, placebo-controlled trial involving 90 patients aged 18 to 65 years, with ASA I or II physical status, scheduled for single-port laparoscopic surgery lasting less than 2 hours. Participants are randomly assigned to either the RSB group or the placebo group, with 45 patients in each group. The RSB group receives bilateral RSB with 15 ml of 0.4% ropivacaine on each side, while the placebo group receives an equal volume of 0.9% saline. The primary outcome is postoperative pain assessed using the Visual Analog Scale (VAS) at multiple time points. Secondary outcomes include opioid consumption, effective activations of the analgesia pump, and postoperative recovery parameters such as time to mobilization and length of hospital stay. The study hypothesizes that preoperative ultrasound-guided bilateral RSB will significantly improve postoperative

DETAILED DESCRIPTION:
Background:

Gynecological single-port laparoscopy has become a preferred surgical approach due to its minimal trauma, concealed scarring, and rapid postoperative recovery. However, postoperative pain and slow recovery of gastrointestinal function remain challenges. Traditional analgesic protocols often rely on opioids, which can cause adverse effects such as nausea, vomiting, bowel paralysis, and respiratory depression.

Objective:

This study aims to evaluate the effects of preoperative ultrasound-guided bilateral rectus sheath block (RSB) on analgesic efficacy and recovery outcomes in patients undergoing gynecological single-port laparoscopy.

Methods:

This is a prospective, randomized, double-blind, placebo-controlled trial. Participants are 90 patients aged 18 to 65 years, ASA I or II, scheduled for single-port laparoscopic surgery lasting less than 2 hours. They are randomly assigned to either the RSB group or the placebo group, with 45 patients in each group. The RSB group receives bilateral RSB with 15 ml of 0.4% ropivacaine on each side, while the placebo group receives an equal volume of 0.9% saline.

Interventions:

RSB Group: Bilateral RSB with 15 ml of 0.4% ropivacaine on each side. Placebo Group: Bilateral injection of 15 ml of 0.9% saline.

Outcome Measures:

Primary Outcome: Postoperative pain assessed using the Visual Analog Scale (VAS) at 30 minutes, 6 hours, 12 hours, and 24 hours postoperatively.

Secondary Outcomes: Opioid consumption, effective activations of the analgesia pump, time to mobilization, time to first passage of flatus, and length of hospital stay.

Hypothesis:

Preoperative ultrasound-guided bilateral RSB will significantly improve postoperative analgesia, reduce opioid consumption, and accelerate postoperative recovery.

Ethics Approval:

The study received approval from the Ethics Committee of Chengdu Jinjiang District Women & Children Health Hospital (approval number: 202214).

Funding:

This study was supported by the Chengdu Medical Research Project (No. 2023465) and the Chengdu Medical Research Project (No. 2022548).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years
* Physical status classified as I or II according to the American Society of Anesthesiologists (ASA)
* Surgical durations of less than 2 hours

Exclusion Criteria:

* Infection at the planned puncture site
* Neurological disorders or nerve injuries
* Conversion to open surgery for various reasons during the procedure
* Coagulation abnormalities

Patients had the option to withdraw from the study at any time if they chose not to continue their participation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is exclusively open to adult females. The study focuses on gynecological single-port laparoscopic procedures, which are medical interventions typically applicable only to women
Enrollment: 90 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Control | 48 hours post-surgery
  ssessment of postoperative pain using the Visual Analog Scale (VAS) scores at multiple time points (30 minutes, 6 hours, 12 hours, 24 hours, and 48 hours after surgery).

SECONDARY OUTCOMES:
Intraoperative Opioid Consumption | Intraoperative
  Total opioid consumption (sufentanil and remifentanil) during the intraoperative period.
Postoperative Recovery Parameters | 24 hours post-surgery
  Time to mobilization,
Postoperative Recovery Parameters | 48 hours post-surgery
  Time to first passage of flatus
Postoperative Recovery Parameters | From postoperative to discharge
  Length of hospital stay
Adverse Event Rates | 48 hours post-surgery
  Incidence of postoperative nausea and vomiting (PONV)
Adverse Event Rates | 48 hours post-surgery
  Incidence of dizziness

CONTACTS AND LOCATIONS:
Overall Officials: Fei Jia, BS, Study Chair — Chengdu Jinjiang District Women & Children Health Hospital
Locations (1):
- Chengdu Jinjiang District Women & Children Health Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
For our study "Effects of Preoperative Bilateral Rectus Sheath Block Guided by Ultrasound on Analgesic Efficacy and Recovery in Gynecological Single-Port Laparoscopy," we have decided not to share Individual Participant Data (IPD). This decision is due to privacy concerns, data security requirements, ethical approval limitations, legal restrictions, and the study's design which did not accommodate data sharing. We believe this aligns with ethical standards and operational capabilities.

REFERENCES:
- [Background] Zhang Y, Zhu Y. Comparison of conventional versus single port laparoscopy for surgical treatment of gynecological diseases: a pilot study. Wideochir Inne Tech Maloinwazyjne. 2022 Mar;17(1):252-260. doi: 10.5114/wiitm.2021.105823. Epub 2021 May 5. PMID 35251414
- [Background] Wang J, Xu X, Xu J. Application of single-port procedure and ERAS management in the laparoscopic myomectomy. BMC Womens Health. 2023 Aug 1;23(1):401. doi: 10.1186/s12905-023-02550-6. PMID 37528370
- [Background] Xu M, Feng Y, Song X, Fu S, Lu X, Lai J, Lu Y, Wang X, Lai R. Combined Ultrasound-Guided Thoracic Paravertebral Nerve Block with Subcostal Transversus Abdominis Plane Block for Analgesia After Total Minimally Invasive Mckeown Esophagectomy: A Randomized, Controlled, and Prospective Study. Pain Ther. 2023 Apr;12(2):475-489. doi: 10.1007/s40122-023-00474-5. Epub 2023 Jan 17. PMID 36648745
- [Background] Liang M, Xv X, Ren C, Yao Y, Gao X. Effect of ultrasound-guided transversus abdominis plane block with rectus sheath block on patients undergoing laparoscopy-assisted radical resection of rectal cancer: a randomized, double-blind, placebo-controlled trial. BMC Anesthesiol. 2021 Mar 24;21(1):89. doi: 10.1186/s12871-021-01295-9. PMID 33761901
- [Background] Chung W, Yoon Y, Kim JW, Kwon SI, Yang JB, Lee KH, Yoo HJ. Comparing two different techniques of rectus sheath block after single port laparoscopic surgery in benign adnexal mass patients: Surgical versus ultrasonography guidance-A randomized, single-blind, case-controlled study. Eur J Obstet Gynecol Reprod Biol. 2017 Oct;217:29-33. doi: 10.1016/j.ejogrb.2017.08.020. Epub 2017 Aug 18. PMID 28843866
- [Background] Mugita M, Kawahara R, Tamai Y, Yamasaki K, Okuno S, Hanada R, Inaoka M, Funato T. Effectiveness of ultrasound-guided transversus abdominis plane block and rectus sheath block in pain control and recovery after gynecological transumbilical single-incision laparoscopic surgery. Clin Exp Obstet Gynecol. 2014;41(6):627-32. PMID 25551952